CLINICAL TRIAL: NCT00806377
Title: Deactivation of Implantable Cardioverter Defibrillator During Non-thoracic Surgical Procedures
Acronym: Dinosur
Status: Completed | Type: Observational
Sponsor: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: EP001
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Implantable Cardioverter-Defibrillators
Keywords: Electromagnetic field; Oversensing; Non-thoracic surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is:

* To document the incidence of electromagnetic oversensing of ICDs during non-thoracic surgery.
* To identify any non-thoracic procedure with a higher incidence of generating electromagnetic oversensing.
* To document the ability of dual chamber ICDs to discriminate electromagnetic oversensing.

DETAILED DESCRIPTION:
Electrocautery devices used during surgery generate a high electromagnetic field with a frequency that may result in ICD oversensing. Oversensing may in turn result in false detection of a ventricular arrhythmia and for the ICD to discharge. Because of this possibility, patients frequently have their ICDs inactivated prior to the procedure.

Although oversensing appears to be highly unlikely in clinical practice, vast resources are utilized in the process of deactivating and reactivating ICDs for surgeries. In addition, there are reports of deaths from failure to reactivate ICDs following elective surgery.

In this study we intend to document the incidence of oversensing, identify procedures with a higher likelihood of oversensing and evaluate the ability of dual chamber ICDs to discriminate electromagnetic oversensing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Medtronic or Boston Scientific single and dual chamber ICDs

Exclusion Criteria:

* Non-thoracic ICD generator placement (abdominal)
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective, non-thoracic surgical procedures will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Electromagnetic oversensing will be reported as a percentage of the total enrolled patients | Assessed at time of procedure

SECONDARY OUTCOMES:
Non-thoracic procedures with a higher incidence of generating electromagnetic oversensing | Assessed at time of procedure
Incidence of dual chamber ICDs discriminating electromagnetic oversensing. | At time of procedure

CONTACTS AND LOCATIONS:
Overall Officials: William T Katsyiannis, MD, Principal Investigator — Minneapolis Heart Institute
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Fiek M, Dorwarth U, Durchlaub I, Janko S, Von Bary C, Steinbeck G, Hoffmann E. Application of radiofrequency energy in surgical and interventional procedures: are there interactions with ICDs? Pacing Clin Electrophysiol. 2004 Mar;27(3):293-8. doi: 10.1111/j.1540-8159.2004.00430.x. PMID 15009852
- [Background] Hauser RG, Kallinen L. Deaths associated with implantable cardioverter defibrillator failure and deactivation reported in the United States Food and Drug Administration Manufacturer and User Facility Device Experience Database. Heart Rhythm. 2004 Oct;1(4):399-405. doi: 10.1016/j.hrthm.2004.05.006. PMID 15851191